CLINICAL TRIAL: NCT07328360
Title: The Efficacy of High-Power Laser Therapy as an Adjunct to Conservative Management in Patients With Meralgia Paresthetica: A Randomized, Assessor-Blinded, Controlled Trial
Brief Title: The Efficacy of High-Power Laser Therapy in Meralgia Paresthetica
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Collaborators: Balikesir University (Other)
Responsible Party: Principal Investigator, Ali Yavuz Karahan, Professor, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AYK&ES&NS
Record Dates: First submitted 2025-12-15; First posted 2026-01-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Meralgia Paresthetica
Keywords: Laser Therapy; Meralgia Paresthetica; Pain; Itching; discopathy
MeSH Terms: conditions — Femoral Neuropathy; Pain; Pruritus

STUDY DESIGN:
Intervention Model Description: Design: A prospective, randomized, assessor-blinded, two-arm parallel-group controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Assessor Blinding: The clinician performing the outcome assessments will be blinded to group allocation.
  Therapist blinding: The therapist applying the laser will not be blinded to the study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: HPLT (Experimental): Application Technique: Scanning technique. The laser probe will be moved slowly and continuously over the entire course of the LFCN (from just medial and inferior to the ASIS, distally along the thigh).
  Interventions: Device: High-power laser; Other: Standard Conservative Care
- Control Group: Sham Laser (Sham Comparator): Identical procedure as Group 1, but with a sham laser applicator that emits no therapeutic energy. The device will beep and display as if it is working.
  Interventions: Other: Sham laser; Other: Standard Conservative Care

INTERVENTIONS:
Device: High-power laser — Operating Mode: Continuous wave Power Output: 10 Watts Energy Dose: A typical effective dose for deep nerves is "800 J per session"
  Arms: Experimental Group: HPLT
Other: Sham laser — The device will beep and display as if it is working.
  Arms: Control Group: Sham Laser
Other: Standard Conservative Care — Education: Advice on avoiding tight belts/trousers, weight loss if applicable, and posture modification.
  -Home Exercise Program: Stretching exercises for the hip flexors (iliopsoas, rectus femoris) and tensor fasciae latae (TFL) to reduce tension on the inguinal ligament.

SUMMARY:
The management of MP typically follows a conservative pathway, encompassing patient education, lifestyle modifications (e.g., avoidance of tight garments, weight loss), pharmacotherapy (such as neuropathic pain agents or corticosteroid injections), and physical therapy. However, evidence supporting the efficacy of these interventions is largely anecdotal or derived from low-quality studies, and a substantial proportion of patients experience persistent symptoms refractory to standard care.

Therefore, the primary objective of this randomized, sham-controlled, assessor-blinded study is to investigate the efficacy of HPLT as an adjunct to standard conservative care on pain intensity, sensory symptoms, and functional capacity in patients with chronic Meralgia Paresthetica. The investigators hypothesize that patients receiving active HPLT will demonstrate significantly greater improvements in these outcomes compared to those receiving a sham laser procedure

DETAILED DESCRIPTION:
Meralgia Paresthetica (MP) is a mononeuropathy characterized by dysesthetic sensations-including burning pain, tingling, and numbness-in the lateral aspect of the thigh. This condition results from the entrapment or compression of the lateral femoral cutaneous nerve (LFCN) as it passes beneath or through the inguinal ligament near the anterior superior iliac spine (ASIS). Common etiological factors include obesity, pregnancy, tight clothing, rapid weight changes, and direct trauma, which increase mechanical stress on the nerve. Despite its relatively high prevalence, MP often remains underdiagnosed and can lead to significant chronic discomfort, functional limitations, and reduced quality of life.

The management of MP typically follows a conservative pathway, encompassing patient education, lifestyle modifications (e.g., avoidance of tight garments, weight loss), pharmacotherapy (such as neuropathic pain agents or corticosteroid injections), and physical therapy. However, evidence supporting the efficacy of these interventions is largely anecdotal or derived from low-quality studies, and a substantial proportion of patients experience persistent symptoms refractory to standard care. For those with intractable pain, invasive procedures like surgical decompression or neurectomy may be considered, though these carry inherent risks of surgical complications and permanent sensory loss. Consequently, there is a pressing need to identify and evaluate novel, effective, and non-invasive therapeutic modalities for MP.

High-Power Laser Therapy (HPLT), also known as high-intensity laser therapy, represents an advanced non-thermal phototherapeutic modality that has gained increasing attention in musculoskeletal and neuropathic pain management. Operating at power outputs typically ranging from 1 to 15 Watts, HPLT utilizes wavelengths (often 980 nm or 1064 nm) that allow for deep tissue penetration. Unlike its low-level counterpart (LLLT), which primarily exerts photobiomodulatory effects, HPLT delivers significant photothermal energy. Its proposed mechanisms of action are multifactorial, including deep tissue analgesia, reduction of inflammation, enhanced microcirculation, and accelerated nerve regeneration. These properties make HPLT a theoretically ideal intervention for entrapment neuropathies like MP, where reducing local inflammation and mechanical stress around the nerve is a primary treatment goal.

Although the application of LLLT for various neuropathies has been explored, the body of literature investigating the specific role of HPLT in compressive mononeuropathies, particularly MP, remains in its infancy. A limited number of studies and case reports have suggested promising analgesic and functional outcomes with HPLT in similar conditions, but robust, randomized controlled trials are lacking.

Therefore, the primary objective of this randomized, sham-controlled, assessor-blinded study is to investigate the efficacy of HPLT as an adjunct to standard conservative care on pain intensity, sensory symptoms, and functional capacity in patients with chronic Meralgia Paresthetica. The investigators hypothesize that patients receiving active HPLT will demonstrate significantly greater improvements in these outcomes compared to those receiving a sham laser procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* Clinical diagnosis of MP (based on history: burning pain, tingling, numbness in the lateral thigh; tenderness over the inguinal ligament near the anterior superior iliac spine (ASIS); and a positive pelvic compression test or Tinel's sign over the lateral femoral cutaneous nerve (LFCN)).
* Symptoms persistent for at least 3 months (chronic).
* A baseline pain intensity of ≥4 on the Numeric Rating Scale (NRS).

Exclusion Criteria:

* Secondary MP (e.g., due to pelvic surgery, trauma, or tumor mass effect confirmed by imaging).
* Significant lumbar radiculopathy (L1-L2).
* Coagulopathy, use of anticoagulants.
* Pregnancy.
* Skin disease or infection in the treatment area.
* Presence of a cardiac pacemaker.
* Severe cognitive impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-07-05 (Estimated); Study Completion 2026-08-05 (Estimated)

PRIMARY OUTCOMES:
PainDETECT | Baseline, 3rd week, 3rd months
  PainDETECT screening questionnaire: PainDETECT is a simple, easy to use screening questionnaire. The questionnaire consists of 9 items and is completed by the patient (no clinical examination is required). There are 7 weighted sensory descriptor items (never to very strongly) and 2 items relating to spatial and temporal pain characteristics. A total score of 19 or more is indicative of likely neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Y Karahan, Prof., Study Chair — University of Usak
Locations (1):
- Usak University, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Authors plan to withhold individual participant data (IPD).